CLINICAL TRIAL: NCT00239421
Title: A Six-Week, Randomized, Double-Blind, Quadruple-Dummy Parallel Group Multiple Dose Study Comparing the Efficacy and Safety of Tiotropium Inhalation Capsules Plus Formoterol Inhalation Capsules to Salmeterol Inhalation Aerosol Plus Fluticasone Inhalation Aerosol in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Six-week Study Comparing the Efficacy and Safety of Tiotropium Plus Formoterol to Salmeterol Plus Fluticasone in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.287
Record Dates: First submitted 2005-10-14; First posted 2005-10-17 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Drug: Test: Tiotropium 18 µg per day (one inhalation capsule) plus 12 µg formoterol twice daily (two times one inhalation capsule)
Drug: Reference: Salmeterol MDI 50 µg (2 puffs of 25 µg each) b.i.d., plus fluticasone propionate MDI 500 µg (2 puffs of 250 µg each) b.i.d.

SUMMARY:
To compare the efficacy and safety of tiotropium plus formoterol in comparison to salmeterol plus fluticasone in COPD patients.

DETAILED DESCRIPTION:
Tiotropium (Spiriva®) is a once-daily inhaled anticholinergic for the treatment of COPD. A six-week, multicentre, randomized, double-blind, parallel group study was conducted to compare the efficacy and safety of the free combination of tiotropium 18 µg once daily plus formoterol 12 µg b.i.d. [Tio+For] to salmeterol 50 µg b.i.d. plus fluticasone 500 µg b.i.d. [Sal+Flu] in COPD patients. Information regarding the differential efficacy and safety of the two different combinations may be essential for physicians to make informed choices of therapy for COPD patients considered candidates for combination therapy.

Following an initial screening visit, subjects entered a two or four-week run-in period in which they received ipratropium (Atrovent®) on a regular basis. At the second visit (Baseline), subjects were randomized into the six-week, double blind portion of the study in which they received either Tio+For or Sal+Flu. After three weeks of treatment, an interim visit was scheduled. After six weeks of treatment, a 12-hour profile of pulmonary function testings (FEV1, FVC) was obtained. Spirometric measurements were performed at pre-dose and 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing. There were two co-primary endpoints: FEV1 area under the curve for the time period 0 to 12 hours (FEV1 AUC0-12) and peak FEV1.

The efficacy evaluation (intention-to-treat) comprised 592 patients [Tio+For: N=297, Sal+Flu: N=295]. The two treatment groups were comparable with regard to demographic data and baseline disease characteristics [Baseline FEV1 (±SE): Tio+For: 1.310 L (±0.026 L); Sal+Flu: 1.325 L (±0.025 L)]. Adjustment was done for baseline and centre-effects.

Study Hypothesis:

The following primary hypotheses (one-sided) were tested with regard to superiority (all means are adjusted means):

H01: FEV1AUC(0-12 hours) (tiotropium+formoterol) <= FEV1AUC (0-12 hours) (salmeterol+fluticasone) versus H11: FEV1AUC(0-12 hours) (tiotropium+formoterol) > FEV1AUC 0-12 hours(salmeterol+fluticasone)

It was stipulated in the protocol that, if the null hypothesis H01 was rejected in favour of H11, then the following hypothesis would be tested:

H01: Peak FEV1 (tiotropium+formoterol) <= Peak FEV1 (salmeterol+fluticasone) versus H11: Peak FEV1 (tiotropium+formoterol) > Peak FEV1 (salmeterol+fluticasone)

Each step was only considered confirmatory providing all previous steps were successful. If any of the previous steps were not successful, any analysis of the current step would have been considered descriptive.

Comparison(s):

Test therapy:

Test product: Tiotropium inhalation capsules plus formoterol inhalation capsules Dose: 18 µg tiotropium per day (one capsule), 12 µg formoterol twice daily (two times one capsule) Mode of administration: inhalation via the Handihaler device (tiotropium), inhalation via the Blue Inhaler device (formoterol)

Reference therapy:

Test product: Salmeterol plus fluticasone propionate Dose: Salmeterol 50 µg (2 puffs of 25 µg each) b.i.d., fluticasone propionate 500 µg (2 puffs of 250 µg each) b.i.d.

Mode of administration: inhalation via MDI

The treatment duration was 42 days each. Primary endpoint measurements were performed on the last treatment day.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent prior to participation in the trial, which includes medication washout and restrictions.
2. All patients must have a diagnosis of chronic obstructive pulmonary disease according to the GOLD criteria and must meet the following spirometric criteria:

   a post-bronchodilator FEV1 < 80% of predicted normal, a post-bronchodilator FEV1/FVC < 70% at Visit 1, and a morning FEV1 <= 65% predicted at Visit 2.
3. Male or female patients 40 years of age or older.
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack-years.
5. Patients must be able to perform technically acceptable pulmonary function tests.
6. Patients must be able to inhale medication in a competent manner from the HandiHaler® device, the Blue Inhaler device, and from a metered dose inhaler (MDI).

Exclusion Criteria:

1. Patients with significant diseases other than COPD.
2. Patients with a recent history (i.e., six months or less) of myocardial infarction.
3. Patients who have been hospitalized for heart failure (NYHA class III or IV) within the past year.
4. Any unstable or life threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year.
5. Patients with a history of cancer within the last five years.
6. Patients with known narrow-angle glaucoma.
7. Patients with a history of asthma, allergic rhinitis or atopy or who have a total blood eosinophil count >= 600/mm3.
8. Patients with a history of life threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis.
9. Patients with known active tuberculosis.
10. Patients with significant alcohol or drug abuse within the past two years.
11. Patients who have undergone thoracotomy with pulmonary resection.
12. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the Screening Visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program that will not be maintained throughout the study.
13. Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy.
14. Patients who are being treated with antihistamines (H1 receptor antagonists) for asthma or excluded allergic conditions.
15. Patients who have taken an investigational drug within one month or six half lives prior to Visit 1.
16. Patients who have been treated with oral beta-adrenergics within one month prior to Visit 1.
17. Patients who have been treated with antileukotrienes or leukotriene receptor antagonists for any disease within one month prior to Visit 1.
18. Patients who have been treated with oral steroids within six weeks prior to Visit 1.
19. Patients who have been treated with monoamine oxidase inhibitors or tricyclic antidepressants within one month prior to Visit 1.
20. Patients who have been treated with cromolyn sodium or nedocromil sodium within one month prior to Visit 1.
21. Patients who have been treated with inhaled steroids within two months prior to Visit 1, including combinations of inhaled steroids and long-acting beta-adrenergics.
22. Patients with known hypersensitivity to anticholinergic drugs, beta adrenergics, lactose or any other components of the inhalation capsule delivery system or any other components of the aerosol delivery systems.
23. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception for the previous three months.
24. Patients with any respiratory infections in the six weeks prior to the Screening Visit (Visit 1) or during the run-in period.
25. Patients who are currently participating in another study.
26. Patients requiring more than eight puffs of salbutamol on three or more consecutive days during the run-in period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605
Dates: Start 2003-11; Primary Completion 2004-09 (Actual); Study Completion 2004-09

PRIMARY OUTCOMES:
The primary efficacy variable was forced expiratory volume in one second (FEV1). There were two co-primary endpoints: FEV1 area under the curve for the time period 0 to 12 hours [FEV1 AUC (0-12)] and peak FEV1 measured after 6 weeks of treatment.

SECONDARY OUTCOMES:
Secondary endpoints were trough FEV1, trough FVC, peak FVC and FVC AUC (0-12) measured at the same times as FEV1 after six weeks of treatment, individual FEV1 and FVC profiles, rescue medication use, peak expiratory flow, results of safety measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (55):
- Austria (3):
  - Med. Uni.-Klinik Graz, Graz
  - Boehringer Ingelheim Investigational Site, Vienna
  - Klinikum Kreuzschwestern Wels, Wels
- Belgium (4):
  - Sint-Vincentius Ziekenhuis, Antwerp
  - CHU Notre Dame des Bruyères, Chênée
  - Heilig Hartziekenhuis Campus Menen, Menen
  - Boehringer Ingelheim Investigational Site, Vosselaar
- Denmark (5):
  - Lungemedicinsk Forskning 2B, Aarhus
  - Bispebjerg Hospital, Copenhagen NV
  - Amtssygehuset i Gentofte, Hellerup
  - Hvidovre Hospital, Hvidovre
  - Odense Universitetshospital, Odense C
- France (5):
  - Centre Hospitalier Germon et Gauthier, Beuvry
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Boehringer Ingelheim Investigational Site, Grenoble
  - Boehringer Ingelheim Investigational Site, Lagord
  - Clinique de la Louvière, Lille
- Germany (16):
  - Boehringer Ingelheim Investigational Site, Berlin
  - MEDARS GmbH, Berlin
  - Klinikum der Ruhr-Universität Bochum, Bochum
  - Klinikum der Universität zu Köln, Cologne
  - ClinGuard GmbH, Dortmund
  - Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - Inamed Research GmbH & Co. KG, Gauting
  - Boehringer Ingelheim Investigational Site, Gelnhausen
  - am Krankenhaus Großhansdorf, Großhansdorf
  - Pneumologisches Forschungsinstitut GmbH, Hamburg
  - Boehringer Ingelheim Investigational Site, Hanover
  - Boehringer Ingelheim Investigational Site, Kiel
  - ClinPharm International GmbH & Co. KG, Leipzig
  - Otto-von-Guericke-Universtität Magdeburg, Magdeburg
  - Boehringer Ingelheim Investigational Site, Minden
  - Boehringer Ingelheim Investigational Site, München
- Netherlands (8):
  - Poli Longziekten, Almelo
  - lokatie Langendijk, Breda
  - Catharina Hospital, Eindhoven
  - Polikliniek Longziekten, Heerlen
  - Poli Longziekten, Hengelo
  - UMC St Radboud ziekenhuis, Nijmegen
  - Sint Franciscus Gasthuis, Rotterdam
  - Afdeling CardioSearch, Veldhoven
- South Africa (10):
  - Tiervlei Trial Centre, Bellville
  - Boehringer Ingelheim Investigational Site, Bloemfontein
  - UCT Lung Institute, Cape Town
  - Boehringer Ingelheim Investigational Site, Cape Town
  - Boehringer Ingelheim Investigational Site, Durban
  - St. Augustine Hospital, Durban
  - QdotPharma, George
  - Boehringer Ingelheim Investigational Site, Johannesburg
  - Boehringer Ingelheim Investigational Site, Paarl
  - Boehringer Ingelheim Investigational Site, Pretoria
- Sweden (4):
  - Lung- och allergikliniken, Länssjukhuset Ryhov, Jönköping
  - Endokrinologmott/Medicinkliniken, Motala
  - Lung och allergikliniken, Stockholm
  - Lung- och allergikliniken, Universitetssjukhuset, Umeå

REFERENCES:
- [Derived] Rabe KF, Timmer W, Sagkriotis A, Viel K. Comparison of a combination of tiotropium plus formoterol to salmeterol plus fluticasone in moderate COPD. Chest. 2008 Aug;134(2):255-262. doi: 10.1378/chest.07-2138. Epub 2008 Apr 10. PMID 18403672